CLINICAL TRIAL: NCT05176275
Title: PET / CT Imaging and Safety of the 68Ga-NOTA-RP25 Molecular Probe in Patients With Lymphoma Who Have Received Prior Therapy Containing CD19 CAR-T Cells
Brief Title: PET / CT Imaging and Safety in Patients With Lymphoma Treated With CD19 Car-t Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Miao Liyan, Chief Pharmacist, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstSoochoowU
Record Dates: First submitted 2021-12-03; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-RP25 (Experimental): Intravenous injection
  Interventions: Diagnostic Test: 68Ga-NOTA-RP25

INTERVENTIONS:
Diagnostic Test: 68Ga-NOTA-RP25 — The proliferation and distribution of CD19 CAR-T cells in lymphoma patients were investigated by PET / CT after injection of 68Ga-NOTA-RP25

SUMMARY:
The proliferation and distribution of CD19 CAR-T cells in lymphoma patients are investigated 68Ga-NOTA-RP25 by PET / CT imaging.

DETAILED DESCRIPTION:
The purpose of this study is to monitor the proliferation and distribution of CD19 CAR-T cells in lymphoma patients by using a novel specific PET tracer 68Ga-NOTA-RP25 for monitoring the proliferation of CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects voluntarily signed the informed consent form and were able to complete the test according to the protocol requirements; 2. Over 18 years old, male or female; 3. Diagnosed as lymphoma and intended to receive CD19 car-t treatment; 4. ECOG score is 0-1; The estimated survival time shall not be less than 3 months;

Exclusion Criteria:

* 1. Participate in other clinical trials other than CAR-T treatment at the same time or within 28 days. If participating in a non intervention clinical trial, it can be included in this study; 2. Patients with a history of allergy; 3. Patients who cannot tolerant PET / CT imaging； 4. Patients who are using anticoagulant drugs or need to use anticoagulant drugs during the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
SUV value of radioactive material uptake in the region of interest | 1 month
  According to the PET / CT imaging results of 68Ga-NOTA-RP25 after iterative reconstruction, PMOD software is used to outline the tumor, brain, liver, heart, tumor and other tissues as regions of interest (ROI)

SECONDARY OUTCOMES:
Safety evaluation index | 1 month
  To observe AE/SAE of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University